CLINICAL TRIAL: NCT01463579
Title: Effectiveness of a Programme of Exercise on Physical Function in Survivors of Critical Illness Following Discharge From the Intensive Care Unit (ICU): a Randomised Controlled Trial
Brief Title: Exercise After Intensive Care Unit: a Randomised Controlled Trial
Acronym: REVIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Brenda O'Neill, Dr Brenda O'Neill, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/0291
Record Dates: First submitted 2011-09-08; First posted 2011-11-02 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Critical Illness; Intensive Care
Keywords: Intensive Care Unit; Critical Illness; Rehabilitation; Exercise Programme
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise programme (Experimental)
  Interventions: Other: Exercise Programme
- Standard Care (Other)
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Exercise Programme — Patients will complete three exercise sessions per week (2 supervised and 1 unsupervised) for 6 weeks. They will receive a written exercise manual which facilitates completion of their exercise programme. The exercise programme will consist of a warm-up, an exercise circuit, a period of aerobic exercise, and a cool down. The programme will be tailored to each patient's ability and needs.
  At the end of the 6 weeks patients will receive a short consultation to set goals relating to continuing exercise at home.
  Arms: Exercise programme
Other: Standard Care — Following ICU admission patients are discharged to hospital wards to the care of a consultant, and the patients are no longer under the care of the ICU team. They are provided with appropriate medical and nursing care, and with referral to other disciplines as necessary. One mobile and able to return home to a carer or another facility they are discharged from hospital. There is usually no support to address potential problems specific to critical illness for patients after ICU discharge.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to test if a 6-week programme of exercise improves physical function and health related quality of life in patients following intensive care who are discharged from hospital. In this study the investigators will compare the physical function and health related quality of life of patients who attend the programme with patients who do not. The 6 week exercise programme will be run by physiotherapy staff, and will mostly take place in a hospital gym. The investigators will measure patients' physical function, exercise capacity, level of breathlessness and their quality of life before and after the 6-week programme, and 6 months later. The investigators will also interview patients to ask their views about the acceptability, enjoyment and satisfaction with the exercise programme. If this study shows that the physical function and health related quality of life are improved in those who took part in the exercise programme, then it will provide useful information which will help the development of services for patients after critical illness. The results will also provide information which will help us design future clinical trials for this patient population.

DETAILED DESCRIPTION:
Most critically ill adult patients require ventilatory support during their intensive care unit stay. Following discharge home patients often still suffer from reduced physical function, exercise capacity, health related quality of life and social functioning for at least 2 years. There is usually no support to address these longer term problems specific to critical illness for patients after hospital discharge. Little research has been carried out into interventions which could improve physical function and quality of life, or enhance speed of recovery in these patients. While there is evidence to support the rehabilitation of critically ill patients within intensive care units, there is a paucity of literature to support rehabilitation following discharge from intensive care and hospital. Therefore, there is a clear and urgent need to investigate interventions which could improve the recovery of patients discharged home after intensive care. This is emerging as a prominent therapeutic objective for the future for this population.

This study will investigate whether a programme of exercise following discharge from hospital will improve outcome in patients following critical illness compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* ICU admission requiring mechanical ventilation > 96 hours
* planned discharge to home (self-care/carer)
* willing and able to participate in exercise
* deemed medically fit to take part in the intervention

Exclusion Criteria:

* declined consent or unable to give consent
* inability to participate due to e.g. any neurological, spinal or skeletal dysfunction affecting ability to exercise
* cognitive impairment affecting ability to understand the intervention or complete questionnaires
* participation in another rehabilitation programme due to ongoing chronic disease
* other medical contraindication to participation in an exercise programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Physical Functioning subscale of the SF-36 | 6 weeks
  The primary outcome measure will be physical function as measured by the physical functioning (PF) subscale of the SF-36v2 following the exercise programme. This is an important outcome that is meaningful to patients. This has been shown to be an acceptable, reliable and valid tool following critical illness.

SECONDARY OUTCOMES:
Physical Functioning Subscale of the SF-36 | 6 months
Rivermead Mobility Index | 6 weeks, 6 months
  Physical Function will also be measured using the Rivermead Mobility Index.
Hand Dynamometry | 6 weeks, 6 months
  Patients have indicated to us that hand function is particularly slow to return after critical illness and that this is important to them. Strength and dexterity will specifically be measured by dynamometry and the Nine Hole Peg Test.
The Nine Hole Peg Test | 6 weeks, 6 months
  Patients have indicated to us that hand function is particularly slow to return after critical illness and that this is important to them. Strength and dexterity will specifically be measured by dynamometry and the Nine Hole Peg Test.
Incremental Shuttle Walk Test | 6 weeks, 6 months
  Exercise capacity will be measured with the Incremental Shuttle Walk Test (ISWT). This is a valid and standardised test of exercise capacity which is responsive to exercise based interventions in other populations. Furthermore the ISWT was used in our pilot study and demonstrated the feasibility and responsiveness of this measure.
Functional Limitations Profile | 6 weeks, 6 months
  Health related quality of life (HRQoL) will also be measured using Functional Limitations Profile (FLP) questionnaire. The FLP questionnaire is a well validated and widely used generic instrument to measure health status in a variety of conditions including critical illness. It provides an estimate of sickness related dysfunction and has both physical and psychosocial dimensions. It was used in our pilot study.
other subscales of the SF-36 | 6 weeks, 6 months
  Health Related Quality of Life (HRQoL) is also assessed using other subscales of the SF-36v2, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores are provided for each of these health domains, and two summary measures of physical and mental health: the Physical Component Summary (PCS) and Mental Component Summary (MCS).
Hospital Anxiety and Depression Scale | 6 weeks, 6 months
  Anxiety and depression function will be measured using the Hospital Anxiety and Depression Scale (HADS). The HADS contains 14 statements and scores from 0-21. Scores of 8-10 indicate the possibility of anxiety or depression, and 11 and above indicate that these are likely to be present. It has been validated in the critical care population.
'Readiness to change' questionnaire | 6 weeks, 6 months
  Patient's readiness to exercise and self efficacy to exercise are important aspects of feasibility when commencing an exercise programme. Readiness to commence exercise following critical illness will be obtained by assessing components relating to the transtheoretical model (stages, processes, decisional balance, self-efficacy). There is evidence of reliability and validity of the questionnaires designed to measure these constructs.
Chronic Disease Self Efficacy Scale (Exercise component) | 6 weeks, 6 months
  The exercise component of the Chronic Disease Self Efficacy Scale will be used to measure self efficacy relating to exercise.
The EuroQol-5D | 6 weeks, 6 months
  The EuroQol-5D is a useful measure of health related quality of life in a mixed critical care population.
Medical Research Council Dyspnoea Scale | 6 weeks, 6 months
  Breathlessness will be measured by the Medical Research Council dyspnoea scale. Breathlessness is a common problem encountered by these patients and an important patient focused outcome.
'Healthcare Utilisation' Questionnaire | 6 months
Semi-structured Interview | 6 months
  Patient's perceptions of the exercise programme will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Brenda O'Neill, PhD, BSc Hons Physiotherapy, Principal Investigator — University of Ulster
Locations (5):
- United Kingdom (5):
  - Northern Health and Social Care Trust, Antrim, Co. Antrim
  - Belfast Health and Social Care Trust, Belfast, Co. Antrim
  - Southern Health and Social Care Trust, Craigavon, Co. Armagh
  - Western Health and Social Care Trust, Londonderry, Co. Londonderry
  - South Eastern Health and Social Care Trust, Dundonald, Co Down

REFERENCES:
- [Background] O'Neill B, McDowell K, Bradley J, Blackwood B, Mullan B, Lavery G, Agus A, Murphy S, Gardner E, McAuley DF. Effectiveness of a programme of exercise on physical function in survivors of critical illness following discharge from the ICU: study protocol for a randomised controlled trial (REVIVE). Trials. 2014 Apr 27;15:146. doi: 10.1186/1745-6215-15-146. PMID 24767671
- [Derived] McDowell K, O'Neill B, Blackwood B, Clarke C, Gardner E, Johnston P, Kelly M, McCaffrey J, Mullan B, Murphy S, Trinder TJ, Lavery G, McAuley DF, Bradley JM. Effectiveness of an exercise programme on physical function in patients discharged from hospital following critical illness: a randomised controlled trial (the REVIVE trial). Thorax. 2017 Jul;72(7):594-595. doi: 10.1136/thoraxjnl-2016-208723. Epub 2016 Nov 15. PMID 27852953